CLINICAL TRIAL: NCT02837835
Title: Comparison of Lung Concentrations of Ceftazidime Administered by Continuous Versus Intermittent Infusion in Patients With Ventilator-associated Pneumonia
Brief Title: Lung Concentrations of Ceftazidime in Patients With Ventilator-associated Pneumonia
Acronym: CEFTALC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104R04
Record Dates: First submitted 2016-07-13; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Ceftazidime

ARMS (2):
- continuous administration of ceftazidime (Experimental)
  Interventions: Drug: ceftazidime
- intermittent administration of ceftazidime (Experimental)
  Interventions: Drug: ceftazidime

INTERVENTIONS:
Drug: ceftazidime — 20 mg/kg of body weight followed by 60 mg/kg/day
  Arms: continuous administration of ceftazidime
Drug: ceftazidime — 20 mg/kg over 30 min every 8 h
  Arms: intermittent administration of ceftazidime

SUMMARY:
Ceftazidime is a beta-lactam compound that exerts a time-dependent bactericidal effect. Numerous arguments are in favor of continuous administration of ceftazidime, both for reasons of clinical efficacy and to preserve bacteriological mutation. The investigators report a prospective, single-center, parallel-group, randomized, controlled trial comparing two modes of administration of ceftazidime, namely, continuous administration (loading dose of 20 mg/kg of body weight followed by 60 mg/kg/day) versus intermittent administration (20 mg/kg over 30 min every 8 h) in 34 patients with ventilator-associated pneumonia due to Gram-negative bacilli. The study was performed over 48 h with 13 and 18 assessments of serum ceftazidime in the continuous-infusion group (group A) and the intermittent-fusion group (group B), respectively. Bronchoalveolar lavage (BAL) was performed at steady state in both groups at 44 h to determine ceftazidime levels in the epithelial lining fluid. The investigators chose a predefined threshold of 20 mg/liter for serum concentrations of ceftazidime because of ecological conditions in our center.

DETAILED DESCRIPTION:
Primary objective

The main objective of this study is to show the continuous administration of superiority ceftazidime versus intermittent administration, in terms of lung tissue concentration of ceftazidime in mechanically ventilated patients with pneumonia caused by a bacillus gram negative.

Methods

Trial

Prospective therapeutic trial in parallel groups, controlled, randomized, single center comparing two methods of administration of ceftazidime (continuous administration by self-pulsed syringe versus discontinuous administration regimens to 3 injections per 24 hours) in patients with severe pneumonia in mechanically ventilated due to gram negative bacillus.

Population

Patients will be enrolled in the Intensive Care Unit of the Reims university hospital.

All patients meeting the inclusion criteria and respecting the criteria of non-inclusions (see below) will be consecutively enrolled in the study after obtaining consent. The allocation of one of the 2 treatment modality will be made by randomization.

Variables and parameters collected in the study:

In addition to sociodemographic variables, variables for inclusion in the study and judgment criteria, different blood and urine tests will be collected:

1. Criteria for inclusion and non-inclusion (see above);
2. Outcome:

   i) concentration in the cell film ceftazidime;

   ii) serum concentration of ceftazidime;

   iii) period during which the serum concentration of ceftazidime is higher than 20 mg/l;
3. Socio-demographic variables: Age, Gender;
4. Blood Assays: Blood gas; Blood Urea, créatinimémie and chemistry panel; serum protein; Complete Blood Count; Beta HCG if women of childbearing age; Liver function tests: AST, ALT, GGT, bilirubin, alkaline phosphatase;
5. Urinary Assays: Creatinine clearance and urinary electrolytes.

ELIGIBILITY:
Inclusion Criteria

* Age >18 years;
* Patients hospitalized in the general intensive care unit of the University Hospital of Reims;
* Nosocomial pneumonia with Gram-negative.

Exclusion Criteria:

* Weight >110 kg;
* Pregnant or breastfeeding women;
* Known allergy to beta - lactam antibiotics;
* Renal impairment: clearance <60 calculated by the Cockcroft and Gault;
* Known history of pulmonary fibrosis;
* Patients included in another research protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
lung tissue concentration of ceftazidime | up to 44 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France

REFERENCES:
- [Result] Cousson J, Floch T, Guillard T, Vernet V, Raclot P, Wolak-Thierry A, Jolly D. Lung concentrations of ceftazidime administered by continuous versus intermittent infusion in patients with ventilator-associated pneumonia. Antimicrob Agents Chemother. 2015 Apr;59(4):1905-9. doi: 10.1128/AAC.04232-14. Epub 2015 Jan 12. PMID 25583727